CLINICAL TRIAL: NCT02791789
Title: Multicenter Pilot Study: Measuring the Evolution of Learning Words and Phrases in Children With Autism Spectrum Disorder Using an Innovative Edutainment Software (SEMATIC)
Brief Title: SEMATIC Pilot Study in Children With Autism Spectrum Disorder Using an Innovative Edutainment Software
Acronym: sematic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 14-HPNCL-10
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; SEMATIC; software
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autism Spectrum Disorder (Other): clinical exam, speech and language therapy and neuropsychological evaluations, Training to the SEMATIC serious game
  Interventions: Other: Autism Spectrum Disorder

INTERVENTIONS:
Other: Autism Spectrum Disorder — Training to the serious game sematic, clinical exam, speech and language therapy and neuropsychological evaluations

SUMMARY:
Use of the software could allow learning of reading code in subjects with ASD through the design of serious games for educational and therapeutic purposes.

This SEMATIC software could improve communication and could be integrated into medical management (speech therapy and neuropsychological).

The benefit of an action research will enable training professionals to autism, cognitive characteristics of autism and the use of IT support for this population.

DETAILED DESCRIPTION:
SEMATIC is an innovative collaborative project which aims to develop an edutainment software for learning words and phrases from logic games. This software is designed for children with autism spectrum disorder (ASD) who do not have the normal prerequisites for learning to read (that is to say: the understanding of words, verbal expression and phonological awareness). In addition, this project is based on hyper competence in the visual field of children with ASD by providing a playful computer support and access to specific visual interests of these children. IT support is a useful tool because it is stable and predictable for focusing the child's attention with ASD. To date, none of learning reading software does exist for children with ASD. This project is based on innovative theoretical and methodological assumptions. These assumptions are derived directly from observation, clinical knowledge of the autistic disorder, testimonies of families and individuals with Asperger Syndrome or Autism High Level and the contributions of the scientific literature in the field of autism.

This software was designed to improve the secondary verbal children with ASD as well as medical care (speech therapist and neuropsychological). The SEMATIC software could be integrated into traditional care for children with ASD. This project is part of an approach of 'action research'. Indeed, this research aims to boost health care teams by training cognitive characteristics of children with ASD and the use of computer support (SEMATIC). Fifteen children with ASD will be recruited in various institutions in the PACA region (departments 06 and 83) to participate in this study. All participants will use the software in the institution where they are usually supported but also at home.

Thus the interest of SEMATIC project is to develop learning words and phrases on computer using logic games to go towards learning the reading code for children with ASD do not have the usual prerequisites. This is a pilot study. There is currently no equivalent method for measuring these changes.

The assessment of learning will be carried out at different times of the protocol. Tests created specifically for the needs of the study will be used. Some tests commonly used in speech therapy and neuropsychological assessments (Standard tools validated on the recommendation of the HAS, 2005) will also be used to include topics and define the characteristics of the population of this study.

ELIGIBILITY:
Inclusion Criteria:

* Review satisfactory medical eligibility criteria
* Diagnosis disorder autism spectrum (ASD) according to the diagnostic criteria of ICD-10 and positive scores to the FA and / or ADOS
* rated severity of autistic symptoms (overall score in the CARS-T scale greater than 30) Non-topics with a functional language (item 11 score ≥ 3 points of the CARS-T)
* a equivalence of higher developmental age or equal to 5 years in analogical reasoning
* n'ayant not develop reading skills by testing the Alouette
* having an interest in visual media (television, computer, touch pad, ...)
* Representatives of parental authority who gave informed written consent
* Subject affiliated to social security

Exclusion Criteria:

* Somatic problems secondarily generate behavioral problems while disrupting their participation in the study
* The Patient having developed reading skills or benefiting from learning to read
* The Patient with no ASD diagnosis according to ICD-10 criteria
* The Patient not affiliated to the social security
* Participant to another research protocol

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
measure learning words and phrases while using SEMATIC in children with ASD and non-readers without functional language | Comparaison between before using SEMATIC serious game and after 11 weeks
  minimum of 50 correct answers out of 100 in the learning score

SECONDARY OUTCOMES:
Evaluate the impact of learning words and phrases on the acquisition of the lexicon (speech and language test ELO) | Comparaison between before using SEMATIC serious game and after 11 weeks
  score to the ELO test
Evaluate the duration of the game necessary to learning | After using SEMATIC serious game after 11 weeks
  score of duration to the ergonomic Questionnaire
Assess the number of sessions necessary to learning | After using SEMATIC serious game after 11 weeks
  score of number of session to the ergonomic Questionnaire
Assess the technical performance and usability of the game platform | After using SEMATIC serious game after 11 weeks
  Ergonomic grid is created and given to parents and educators to evaluate the software, usability and technical performance of the game
Evaluate the satisfaction of organizing the SEMATIC survey of parents and educators | After using SEMATIC serious game after 11 weeks
  score to the satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie SERRET, MD, Principal Investigator — Fondation Lenval - Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (1):
- Fondation LENVAL - Hôpitaux Pédiatriques de Nice CHU-LENVAL, Nice, France

IPD SHARING:
Plan to Share IPD: No